CLINICAL TRIAL: NCT04827667
Title: Impact of PD1-lymphocytes in Bronchoalveolar Lavage of Patients With Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Daniela Gompelmann, Prof. Dr. med., University of Vienna
Other Study IDs: Version 1 20.04.2020
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with lung cancer: In lung cancer patients with indication for bronchoscopy, bronchoalveolar lavage is performed to assess PD1-lymphocytes.
  Interventions: Diagnostic Test: bronchoalveolar lavage
- Patients wiht interstitial lung disease: In patients with interstitial lung disease with indication for bronchoscopy, bronchoalveolar lavage is performed to assess PD1-lymphocytes.
  Interventions: Diagnostic Test: bronchoalveolar lavage
- Patients with asthma: In patients with asthma with indication for bronchoscopy, bronchoalveolar lavage is performed to assess PD1-lymphocytes.
  Interventions: Diagnostic Test: bronchoalveolar lavage

INTERVENTIONS:
Diagnostic Test: bronchoalveolar lavage — Bronchoalveolar lavage is performed by instillation and suction of saline in the middle lobe during bronchoscopy. Cytological examination and flow cytometry will be performed to assess PD-1lymphoctes.

SUMMARY:
The aim of this trial is to assess PD1-lymphocytes in bronchoalveolar lavage in patients with lung cancer, ILD and asthma.

DETAILED DESCRIPTION:
In this trial, 20 patients with lung cancer, 10 patients with asthma and 10 patients with interstitial lung disease who have to undergo bronchocospy for medical reasons are enrolled. In each patient, bronchoalveolar lavage is performed to assess PD1-lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* patients with lung cancer, asthma or ILD and indication for bronchoscopy for medical reasons
* Ability to provide informed consent

Exclusion Criteria:

* acute excacerbation in patients with asthma or ILD
* endoluminal tumor growth or penumonia in patients with lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or proven lung cancer, asthma or instertitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess and compare PD1-lmyphocytes in bronchoalveolar lavage in patients with malignant and benign lung diseases to evluate their impact in lung cancer patients | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided